CLINICAL TRIAL: NCT00003600
Title: A Phase III Randomized Double-Blind Study of Erythropoietin Versus Placebo in Anemic Patients With Cancer Undergoing Chemotherapy
Brief Title: Epoetin Alfa in Treating Anemia in Patients Who Are Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-979253; CDR0000066673 (Registry Identifier: PDQ (Physician Data Query)); NCI-P98-0133
Record Dates: First submitted 1999-11-01; First posted 2004-02-20 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Anemia; Breast Cancer; Chronic Myeloproliferative Disorders; Drug/Agent Toxicity by Tissue/Organ; Leukemia; Lung Cancer; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Precancerous Condition; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Anemia; Breast Neoplasms; Myeloproliferative Disorders; Drug-Related Side Effects and Adverse Reactions; Leukemia; Lung Neoplasms; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Precancerous Conditions | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- epoetin alfa (Experimental): Patients receiving chemotherapy are randomized to receive epoetin alfa subcutaneously once a week for a maximum of 16 weeks Quality of life is assessed at randomization and monthly throughout study. Patients are followed every 6 months for 1 year.
  Interventions: Biological: epoetin alfa
- placebo (Placebo Comparator): Patients receiving chemotherapy are randomized to receive placebo subcutaneously once a week for a maximum of 16 weeks. Quality of life is assessed at randomization and monthly throughout study. Patients are followed every 6 months for 1 year.
  Interventions: Other: placebo

INTERVENTIONS:
Biological: epoetin alfa
  Arms: epoetin alfa
Other: placebo
  Arms: placebo

SUMMARY:
RATIONALE: Epoetin alfa may stimulate red blood cell production and treat anemia in patients with cancer who are receiving chemotherapy. It is not yet known whether epoetin alfa is more effective than a placebo in treating anemia in patients receiving chemotherapy.

PURPOSE: Randomized double blinded phase III trial to compare the effectiveness of epoetin alfa with a placebo in treating anemia in cancer patients who are receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether epoetin alfa treatment improves the quality of life in anemic patients who are undergoing chemotherapy for advanced malignancy. II. Determine whether epoetin alfa increases hemoglobin levels and decreases transfusion requirements in these patients. III. Validate or refute the use of an algorithm using pre- and posttreatment epoetin alfa, ferritin, and hemoglobin levels to predict 16 weeks response or no response to therapeutic doses of epoetin alfa as set forth by these patients. IV. Explore whether anemic patients receiving platinum-containing chemotherapy regimens experience less nephrotoxicity if they receive concurrent epoetin alfa compared to those who receive placebo.

OUTLINE: This is a randomized, double blind study. Patients are stratified by primary malignant disease (lung vs breast vs other), life expectancy (4-6 months vs greater than 6 months), planned concurrent radiotherapy (yes vs no), and degree of anemia (mild or at least 9 g/dL vs severe or less than 9 g/dL). Patients receiving chemotherapy are randomized to receive epoetin alfa subcutaneously once a week for a maximum of 16 weeks (arm I) or placebo subcutaneously once a week for a maximum of 16 weeks (arm II). Quality of life is assessed at randomization and monthly throughout study. Patients are followed every 6 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Anemic: Hemoglobin in males less than 11.5 g/dL; hemoglobin in females less than 10.0 g/dL No anemia secondary to B12, folic acid, or iron deficiency No anemia secondary to gastrointestinal bleed or hemolysis No anemia secondary to a primary or chemotherapy-induced myelodysplastic syndrome No anemia secondary to acute lymphocytic leukemia Histologically confirmed advanced malignancy Lung Breast Other Currently receiving myelosuppressive, cytotoxic chemotherapy for advanced cancer No patients receiving adjuvant therapy for cancer that has been surgically removed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: At least 4 months Hematopoietic: See Disease Characteristics Hepatic: Not specified Renal: Not specified Cardiovascular: No uncontrolled hypertension (systolic at least 180, diastolic at least 100) Other: Normal or elevated ferritin No known hypersensitivity to epoetin alfa Must be able to reliably take oral medication Must be alert and mentally competent Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 1 year since prior epoetin alfa At least 2 weeks since prior red blood cell transfusions No concurrent peripheral blood stem cell or bone marrow transplantation Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Concurrent radiotherapy allowed Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 1998-12; Primary Completion 2001-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Quality of life | Up to 12 months

SECONDARY OUTCOMES:
Predict response | Up to 12 months
Response rate | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Witzig, MD, Study Chair — Mayo Clinic
Locations (21):
- United States (20):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Howard University Cancer Center, Washington D.C., District of Columbia
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada